CLINICAL TRIAL: NCT04268784
Title: A Phase 1, Single-Center, Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of DNL343 In Healthy Volunteers
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of DNL343 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Denali Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: DNLI-F-0001; 2019-004027-21 (EudraCT Number)
Record Dates: First submitted 2020-02-10; First posted 2020-02-13 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DNL343 (Experimental): Cohort A: Single-ascending dose; Cohort B: Multiple-ascending doses
  Interventions: Drug: DNL343
- Placebo (Placebo Comparator): Cohort A: Single-ascending dose; Cohort B: Multiple-ascending doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DNL343 — Single and repeating oral dose(s)
  Arms: DNL343
Drug: Placebo — Single and repeating oral dose(s)
  Arms: Placebo

SUMMARY:
This is a Phase 1 study carried out at a single site in 88 healthy male subjects and healthy female subjects of non childbearing potential to investigate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of DNL343.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Women of non-childbearing potential and men; aged 18-50 years, inclusive
* BMI 18-32 kg/m², inclusive, and body weight of at least 50 kg

Key Exclusion Criteria:

* History of clinically significant neurologic, psychiatric, endocrine, pulmonary, cardiovascular, gastrointestinal, hepatic, pancreatic, renal, metabolic, hematologic, immunologic, or allergic disease, or other major disorders

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) including serious adverse events (SAEs), and discontinuations due to TEAEs | Up to 20 days
PK parameter: The area under the concentration-time curve from time zero extrapolated to infinity (AUC0-∞) of DNL343 in plasma | Up to 20 days
PK parameter: The area under the concentration-time curve from zero to 12 or 24 hours for twice daily (BID) or once daily (QD) dosing, respectively (AUC0-τ) of DNL343 in plasma | Up to 20 days
PK parameter: Maximum observed concentration (Cmax) of DNL343 in plasma | Up to 20 days
PK parameter: Area under the concentration-time curve from time zero to the time of last quantifiable concentration (AUC[0-last]) of DNL343 in plasma | Up to 20 days
PK parameter: Time to maximum observed concentration (Tmax) of DNL343 in plasma | Up to 20 days
PK parameter: Apparent terminal elimination rate constant (λz) with the respective t½ of DNL343 in plasma | Up to 20 days

SECONDARY OUTCOMES:
PK parameter: The amount of DNL343 excreted in urine from time zero to 48 hours postdose (Ae48) | Up to 20 days
PK parameter: Estimation of renal clearance (CLR) | Up to 20 days
PK parameter: Concentration of DNL343 in cerebrospinal fluid (CSF) | Up to 20 days
The PD of DNL343 in blood as measured by percent reduction of integrated stress response (ISR) protein levels measured by enzyme-linked immunosorbent assay (ELISA) | Up to 20 days
The PD of DNL343 in blood as measured by percent reduction in ISR gene expression levels measured by quantitative polymerase chain reaction (qPCR) | Up to 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard Tsai, MD, Study Director — Denali Therapeutics Inc.
Locations (1):
- Centre for Human Drug Research (CHDR), Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No